CLINICAL TRIAL: NCT07355166
Title: Suzetrigine Versus Usual-care Opioids for Postoperative Pain After Common Ambulatory Orthopaedic Sports Procedures - A Randomized Control Trial
Brief Title: Suzetrigine Versus Usual-care Opioids for Postop Pain in Sports
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jomar Aryee, Orthopaedic Sports Fellow, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-25-2108
Record Dates: First submitted 2026-01-01; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain Management
Keywords: Suzetrigine; Journavx; Opioid Use; ACL Reconstruction; Rotator Cuff Repair; Postoperative Pain Management

STUDY DESIGN:
Masking Description: Statistical Analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suzetrigine Arm (Experimental): Patients in both groups will receive a common multimodal pain control regimen which includes a preoperative regional anesthesia, a 14-day supply of 1000mg acetaminophen BID, and a 14-day supply of 500mg naproxen BID. Patients randomized to the Suzetrigine arm will receive a loading dose of Suzetrigine 100mg in PACU postoperatively and a 7-day supply of 50mg suzetrigine BID for 1 week total.
  Patients in this group will also receive 25 tablets of 5mg of oxycodone for rescue pain control.
  Interventions: Drug: Suzetrigine
- Opioid Arm (Experimental): Patients in both groups will receive a common multimodal pain control regimen which includes a preoperative regional anesthesia, a 14-day supply of 1000mg acetaminophen BID, and a 14-day supply of 500mg naproxen BID. Patients randomized to the Opioid arm will also receive 25 tablets of 5mg of oxycodone and will not receive a Suzetrigine prescription.
  Interventions: Drug: Multimodal Pain Regimen

INTERVENTIONS:
Drug: Suzetrigine — Patients in this group will receive a preoperative regional anesthesia block, a 14-day supply of 1000mg acetaminophen BID, a 14-day supply of 500mg naproxen BID, a loading dose of Suzetrigine 100mg in PACU postoperatively, a 7-day supply of 50mg suzetrigine BID and 25 tablets of 5mg of oxycodone for rescue pain control postoperatively.
  Other Names: Journavx
  Arms: Suzetrigine Arm
Drug: Multimodal Pain Regimen — Patients in this group will receive a preoperative regional anesthesia block, a 14-day supply of 1000mg acetaminophen BID, a 14-day supply of 500mg naproxen BID, and 25 tablets of 5mg of oxycodone for PRN pain control postoperatively.
  Arms: Opioid Arm

SUMMARY:
The goal of this clinical trial is to learn if a Suzetrigine-based multimodal pain regimen can reduce the volume of opioid consumption while maintaining non-inferior pain control compared to an opioid-based multimodal pain regimen after common ambulatory orthopaedic sports procedures. The main questions it aims to answer are:

1. Does including Suzetrigine in the multimodal pain regimen lower the volume of opioids consumed by participants while maintaining non-inferior pain control?
2. How does the side-effect profile of a Suzetrigine-based multimodal postop pain regimen compare to that of an opioid-based multimodal postoperative pain regimen?

Eligible participants will be assigned to receive one of the postop pain regimens and report their opioid use, their pain level, and the side effects they faced every day for 7 days.

DETAILED DESCRIPTION:
Pain control after most arthroscopic and open orthopaedic sports surgeries in the ambulatory setting is dependent on multimodal pain regimens that include the use of narcotics. These medications are often considered necessary for appropriate pain control but pose risks of harm to patients through systemic side effects, potential for overdose, and potential for long-term dependence. They also pose risks to society through diversion, fueling the economically burdensome opioid crisis, and being a nidus for drug-related crimes. Suzetrigine (Journavx) was FDA-approved in January of 2025 for use in the management of acute pain. It is the first non-opioid analgesic approved since celecoxib (anti-inflammatory) in the late 1990's and has been shown to provide non-inferior pain control when compared to placebo as well as to opioid-based drug regimens in some postoperative settings. It's efficacy in reducing postoperative opioid exposure without sacrificing pain control after common ambulatory orthopaedic sports procedures that already use multimodal/regional anesthesia has yet to be studied in a controlled fashion.

At the University of Califronia Los Angeles (UCLA), multimodal strategies for patients undergoing common ambulatory orthopaedic sports procedures like primary ACL reconstruction or rotator cuff repair currently include regional anesthesia, acetaminophen, NSAIDs, and opioids. Since FDA approval, Suzetrigine has been incorporated into postoperative pain management at UCLA for select patients, but has not been uniformly adopted. Evaluating its role in a controlled, randomized setting among patients undergoing common ambulatory Orthopaedic sports procedures will provide important data on best practices when incorporating it within current multimodal protocols as well as its impact on postoperative opioid use in these settings.

This study aims to evaluate its efficacy and opioid-sparing potential in patients undergoing an archetypal outpatient, Orthopaedic sports knee procedure - primary ACL reconstruction - and to inform its potential integration into enhanced recovery pathways.

This aim will be achieved by investigating whether a Suzetrigine based multimodal regimen affects total opioid consumption over 7 days after surgery when compared to an opioid-based multimodal regimen, while maintaining non-inferior pain control at 48 hours

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing reconstruction of primary ACL tear

Exclusion Criteria:

* Concurrent ligamentous injuries requiring surgical intervention
* Full thickness cartilage injury requiring discrete surgical intervention
* Chronic opioid use
* Significant hepatic disease (Child/Pugh C)
* Women who are pregnant or breastfeeding
* Women of childbearing age using hormonal contraceptives containing progestins other than levonorgestrel and norethindrone
* Allergies or intolerance to any study medications
* Inability to complete ePROs (due to literacy or infirmity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
7-Day MME Consumption | 7 days
  Total opioids consumed by patients measured in morphine milliequivalents for the first seven days postoperatively

SECONDARY OUTCOMES:
SPID-48 | 48 hours
  Time-weighted Sum of Pain Intensity Difference over 48 hours used to quantify pain relief by summing a patient's pain reduction from their baseline score over a 48-hour period.
7-Day Opioid Free Rate | 7 days
  The percentage of patients who avoid opioid use after medical procedures
Opioid Side Effect Rate | 7 days
  Proportion of patients reporting instances of nausea, constipation, dizziness, or loss of appetite
Suzetrigine Side Effect Rate | 7 Days
  Proportion of patients reporting muscle aches, muscle spasm, or itchiness

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones J, Correll DJ, Lechner SM, Jazic I, Miao X, Shaw D, Simard C, Osteen JD, Hare B, Beaton A, Bertoch T, Buvanendran A, Habib AS, Pizzi LJ, Pollak RA, Weiner SG, Bozic C, Negulescu P, White PF; VX21-548-101 and VX21-548-102 Trial Groups. Selective Inhibition of NaV1.8 with VX-548 for Acute Pain. N Engl J Med. 2023 Aug 3;389(5):393-405. doi: 10.1056/NEJMoa2209870. PMID 37530822